CLINICAL TRIAL: NCT01822769
Title: Cardiopulmonary Rehabilitation for Adolescents and Adults With Congenital Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Alexander Opotowsky, Assistant Professor, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P00005391
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Congenital Heart Disease; Heart Defects, Congenital
Keywords: congenital heart disease; adult congenital heart disease; cardiac rehabilitation; cardiopulmonary rehabilitation; exercise; cardiopulmonary exercise testing; peak vO2; quality of life
MeSH Terms: conditions — Heart Defects, Congenital; Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cardiopulmonary rehabilitation (Experimental): The subjects will attend 2 sessions each week for 12 weeks. Each session will be approximately 2 hours in duration, consisting of both exercise (aerobic and strength,~60 minutes) and education. In addition, subjects will be directed to participate in 3 weekly ~40 minute home exercise training sessions, personalized to their level of aerobic conditioning.
  Interventions: Other: Cardiopulmonary rehabilitation
- Standard of care (Other): Subjects randomized to standard of care will not be enrolled in a rehabilitation program, but may receive any other clinically indicated exercise training or other intervention (e.g., an exercise prescription).
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Cardiopulmonary rehabilitation — See Arm Description
  Arms: Cardiopulmonary rehabilitation
Other: Standard of care — See Arm Description
  Arms: Standard of care

SUMMARY:
The hypothesis of this study is that participation in a formal cardiopulmonary rehabilitation program improves aerobic exercise capacity and quality of life over the medium term for patients with congenital heart disease with reduced exercise capacity. To test this hypothesis, subjects will be randomized to either receive a 12-week cardiopulmonary rehabilitation program or standard of care, with interval testing of aerobic capacity and other physiologic markers improved fitness, as well as assessment of quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to participate in a 12-week cardiac rehabilitation program and repeated cardiopulmonary exercise testing
* pVO2≤80% predicted (impaired aerobic capacity) on baseline exercise test
* congenital heart disease of at least moderate complexity

Exclusion Criteria:

* Cardiac intervention (cath/surg) within prior 6m
* Planned cardiac intervention (cath/surg) within 12m
* Formal cardiac rehabilitation within 24m
* Current/recent (delivery<90d prior) pregnancy, planned pregnancy within 12m
* Active heart failure, hospitalization or major change in clinical status over prior 30d
* Other recent or planned events expected to have a significant impact on exercise capacity
* Baseline oxygen saturation <92%

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in aerobic exercise capacity (peak VO2) | Baseline to 3 months (primary)

SECONDARY OUTCOMES:
Change in quality of life measurement | Baseline to 3 months (primary)

OTHER OUTCOMES:
Change in peak cardiac output and its components (SV/HR) | Baseline to 3 months (primary)
Mechanism of change in peak VO2 | Baseline to 3 months (primary)
  Cardiac output will be assessed and O2 delivery/extraction will be estimated to define mechanisms of improvement in exercise capacity.
Change in ventilatory efficiency | Baseline to 3 months (primary)
Change in strength (dynamometry) | Baseline to 3 months (primary)
Change in pulse wave velocity | Baseline to 3 months
Change in circulating biomarkers | Baseline to 3 months (primary)
Change in markers of pulse reflection | Baseline to 3 months
Incidence of arrhythmia and other adverse events during cardiopulmonary rehabilitation | Baseline to 3 months
Change in physical activity | Baseline to 3 months
  Survey and accelerometry
Change in markers of ventricular function | Baseline to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Opotowsky, Principal Investigator — Boston Children's Hospital, Brigham and Women's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States